CLINICAL TRIAL: NCT05965427
Title: Morbidity, Mortality And Risk Factors of Mpox in HIV Negative High Risk Sexual Health Clinic Attenders and People Living With HIV
Acronym: MASH1
Status: Completed | Type: Observational
Sponsor: NEAT ID Foundation (Other)
Collaborators: European Commission (Other); PENTA Foundation (Network)
Responsible Party: Sponsor
Other Study IDs: 606
Record Dates: First submitted 2023-06-23; First posted 2023-07-28 (Actual); Results first posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-07

CONDITIONS: Monkeypox; HIV Coinfection
MeSH Terms: conditions — Mpox, Monkeypox; HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PLWHIV and Mpox coinfection: People living with HIV(PLWHIV) who are at least 18 years of age, with confirmed Mpox infection by documented, positive result on PCR testing of lesions from 1st May 2022 to 1st December 2023.
  Interventions: Other: No intervention
- HIV negative PrEP users with Mpox infection: HIV negative PrEP (Pre-exposure prophylaxis) users who are at least 18 years of age, with confirmed Mpox infection by documented, positive result on PCR testing of lesions from 1st May 2022 to 1st December 2023.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Study is retrospective data collection only

SUMMARY:
This data collection study aims to describe and compare the outcomes of Mpox on people living with HIV (PLHIV) and HIV-negative individuals who are on pre-exposure prophylaxis (PrEP). The study also aims to identify risk factors for specific Mpox outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MPX was more than 90 days prior to data collection
* Confirmed MPX infection by documented PCR testing of lesions between 1st May 2022 to 1st December 2023
* At least 18 years of age
* Cases (PLWHIV + MPX) i) Documented HIV-1 infection
* Cases (PrEP users + MPX) i) Attended a clinic to receive PrEP

Exclusion Criteria:

* MPX diagnosed based on clinical criteria only
* MPX diagnosis was within the last 90 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People living with HIV who are currently sexually active and HIV negative high-risk Sexual Health Clinic attenders (PrEP users) with Mpox
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-05-07 (Actual); Study Completion 2025-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolo Girometti, MD, Principal Investigator — Chelsea and Westminster NHS Trust
Locations (9):
- France (2):
  - Hôpital Bichat Claude Bernard, Paris
  - Hôpital Pitié-Salpêtrière, Paris
- Euroguidelines, Warsaw, Poland
- Spain (5):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitari Germans Trias I Pujol, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital San Carlos, Madrid
  - Hospital Universitario La Paz, Madrid
- Chelsea and Westminster Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Deidentified real-world retrospective, routine data was collected PLWHIV (people living with HIV) who are currently sexually active and HIV negative high-risk Sexual Health Clinic attenders (PrEP users) with Mpox at clinical sites in the UK and Europe.
Pre-assignment Details: This is observational retrospective cohort data collection study. Data was collected from adult PrEP users and PLWHIV with confirmed mpox infection by documented, positive result on PCR testing of lesions from 1st May 2022 to 1st December 2023, at least 90 days prior to data collection.
Groups:
- PLHIV and Mpox Coinfection; HIV Negative PrEP Users With Mpox Infection: No intervention: Study is retrospective data collection only
Period: Overall Study
Arm/Group | PLHIV and Mpox Coinfection | HIV Negative PrEP Users With Mpox Infection
Started | 946 | 1054
Completed | 946 | 1054
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PLWHIV and Mpox Coinfection | HIV Negative PrEP Users With Mpox Infection | Total
Number analyzed (Participants) | 946 | 1054 | 2000
Age, Customized [Count of Participants; unit: Participants]
  Age Category : <30 | 108 | 209 | 317
  Age Category : 30-40 | 433 | 521 | 954
  Age Category : >40 | 405 | 324 | 729
Sex/Gender, Customized [Number; unit: participants]
  Sex/Gender : Male sex at birth | 946 | 1054 | 2000
  Sex/Gender : Male gender identity | 922 | 1040 | 1962
  Sex/Gender : Female gender identity | 24 | 12 | 36
  Sex/Gender : Non-binary | 0 | 2 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 282 | 445 | 727
  Mixed or multiple | 42 | 32 | 74
  Black | 29 | 28 | 57
  Asian | 8 | 35 | 43
  Other | 28 | 49 | 77
  Not stated | 557 | 465 | 1022
Region of Enrollment [Number; unit: participants]
  Poland | 67 | 19 | 86
  United Kingdom | 250 | 521 | 771
  France | 104 | 156 | 260
  Spain | 525 | 358 | 883
Orthopoxvirus vaccination [Count of Participants; unit: Participants] — The number of participants who had previously received an Orthopoxvirus vaccine Population: Vaccination history was not available for all participants.
  Participants
    number analyzed (Participants) | 562 | 431 | 993
    (all) | 82 | 51 | 133
Comorbidities [Count of Participants; unit: Participants] — The number of participants with comorbidities were collected where available. Other category includes history of myocardial infarction, congestive heart failure, peripheral vascular disease, stroke or ischemic attack, dementia, chronic obstructive pulmonary disease, history of pneumonia, connective tissue disease, peptic ulcer disease, hemiplegia, paralysis of arm(s) or leg(s), current or history of cancer (excluding lymphoma). Immunosuppression is defined as presence of either leukaemia or lymphoma or significant CD4 count depletion (either CD4 count <200/mm3 and/or CD4% <10%)] Population: Due to the retrospective data collection nature of this study, data on comorbidities were not available for all participants.
  Participants
    Liver disease: number analyzed (Participants) | 934 | 1048 | 1982
    Liver disease | 35 | 3 | 38
    Chronic kidney disease: number analyzed (Participants) | 931 | 1048 | 1979
    Chronic kidney disease | 3 | 1 | 4
    Diabetes: number analyzed (Participants) | 929 | 1048 | 1977
    Diabetes | 8 | 1 | 9
    Lymphoma or leukaemia: number analyzed (Participants) | 934 | 1048 | 1982
    Lymphoma or leukaemia | 11 | 2 | 13
    AIDS defining condition: number analyzed (Participants) | 935 | 1049 | 1984
    AIDS defining condition | 316 | 0 | 316
    Mental health condition: number analyzed (Participants) | 928 | 1017 | 1945
    Mental health condition | 66 | 39 | 105
    Immunosuppressed: number analyzed (Participants) | 822 | 1048 | 1870
    Immunosuppressed | 101 | 2 | 103
    Other: number analyzed (Participants) | 932 | 1048 | 1980
    Other | 44 | 18 | 62
Sexual history [Count of Participants; unit: Participants] — Recent sexual history (3 months)
  Participants
    Multiple sexual partners | 523 | 743 | 1266
    Any recent or concurrent sexually transmitted infection | 335 | 373 | 708
HIV status [Mean (Standard Deviation); unit: years] — Time since HIV diagnosis at mpox diagnosis Population: This measure is only applicable to the PLWHIV cohort, therefore no data was collected for the HIV-negative PrEP users cohort.
  years
    number analyzed (Participants) | 946 | 0 | 946
    (all) | 9.5 (6.6) |  | 9.5 (6.6)
Antiretroviral Therapy [Count of Participants; unit: Participants] — The number of participants in the PLWHIV cohort receiving antiretroviral therapy/treatment (ART). Population: This measure is only applicable to the PLWHIV cohort, therefore no data was collected for the HIV-negative PrEP users cohort. ART variables were not available for one individual in the PLWHIV cohort so this participant is excluded from the analysis.
  Participants
    Currently receiving ART: number analyzed (Participants) | 945 | 0 | 945
    Currently receiving ART | 925 |  | 925
    Not currently receiving ART: number analyzed (Participants) | 945 | 0 | 945
    Not currently receiving ART | 20 |  | 20
CD4 count [Mean (Standard Deviation); unit: cells/mm^3] — Last CD4 count before mpox diagnosis Population: This measure is only applicable to the PLWHIV cohort, therefore no data was collected for the HIV-negative PrEP users cohort. CD4 data was not available for all participants in the PLHIV cohort and was collected where available.
  cells/mm^3
    number analyzed (Participants) | 824 | 0 | 824
    (all) | 677 (357) |  | 677 (357)
HIV RNA levels [Mean (Standard Deviation); unit: copies/ml] — Most recent HIV RNA levels before mpox diagnosis Population: This measure is only applicable to the PLWHIV cohort, therefore no data was collected for the HIV-negative PrEP users cohort. HIV RNA data was not available for all participants in the PLHIV cohort and was collected where available.
  copies/ml
    number analyzed (Participants) | 846 | 0 | 846
    (all) | 7673 (59693) |  | 7673 (59693)
HIV RNA level <50 copies/mL [Count of Participants; unit: Participants] — The number of participants with HIV RNA <50 copies/mL Population: This measure is only applicable to the PLWHIV cohort, therefore no data was collected for the HIV-negative PrEP users cohort. HIV RNA data was not available for all participants in the PLHIV cohort and was collected where available.
  Participants
    number analyzed (Participants) | 846 | 0 | 846
    (all) | 755 |  | 755

OUTCOME MEASURES:

1. Primary Outcome: Severe Mpox Lesions
Description: The number of participants with severe Mpox lesions. Severity of lesions will be assessed by the peak number of lesions and peak number of sites. Participants with ≥100 lesions at peak severity will be classified as having "severe lesions".
Time Frame: From date of disease onset (first symptom) until date of peak number of lesions and sites recorded (up to 3 months)
Population: Skin lesion severity could not be analysed for all participants as the number of lesions were not available due to the retrospective data collection nature of this study.
Measure: Number; unit: participants
Groups:
- PLWHIV and Mpox Coinfection: People living with HIV (PLWHIV) who are at least 18 years of age, with confirmed MPX infection by documented, positive result on PCR testing of lesions from 1st May 2022 to 1st December 2023.
- HIV Negative PrEP Users With Mpox Infection: PrEP (Pre-exposure prophylaxis) users who are at least 18 years of age, with confirmed MPX infection by documented, positive result on PCR testing of lesions from 1st May 2022 to 1st December 2023.
Arm/Group | PLWHIV and Mpox Coinfection | HIV Negative PrEP Users With Mpox Infection
Number analyzed (Participants) | 766 | 906
participants | 6 | 2
Statistical Analysis 1: Comparison: PLWHIV and Mpox Coinfection vs HIV Negative PrEP Users With Mpox Infection; Test type: Superiority; p = 0.097, Chi-squared

2. Primary Outcome: Clinical Complications Associated With Mpox
Description: Complications which will be collected are as follows:
  * Severe rectal and/or perianal pain (i.e. due to perianal/anal abscess, proctitis)
  * Tonsillitis and/or dysphagia
  * Secondary bacterial infection on affected skin
  * Urological complications (genital oedema, urinary retention)
  * Ocular involvement (conjunctivitis, corneal involvement, periorbital cellulitis)
  * Central nervous system involvement (encephalitis, meningitis, focal neurology signs)
  * Pneumonia/pulmonary abscess or necrotizing involvement
  * Myocarditis
  * Diarrhoea
  A composite outcome representing the presence of any specified clinical complication will be analysed. This composite outcome will be derived by identifying participants who have experienced one or more of the listed clinical complications during the observation period.
Time Frame: From date of disease onset (first symptom) until date of clinical resolution e.g. lesion resolution, hospital discharge or death (up to 3 months)
Population: Clinical complication data was not available for available for all participants due to the retrospective data collection nature of this study.
Measure: Count of Participants; unit: Participants
Arm/Group | PLWHIV and Mpox Coinfection | HIV Negative PrEP Users With Mpox Infection
Number analyzed (Participants) | 938 | 1051
Participants
  Severe rectal and/or perianal pain: number analyzed (Participants) | 938 | 1049
  Severe rectal and/or perianal pain | 192 | 242
  Tonsilitis: number analyzed (Participants) | 938 | 1050
  Tonsilitis | 38 | 50
  Dysphagia: number analyzed (Participants) | 937 | 1051
  Dysphagia | 21 | 22
  Secondary bacterial infection on affected skin: number analyzed (Participants) | 937 | 1049
  Secondary bacterial infection on affected skin | 108 | 124
  Urological complications: number analyzed (Participants) | 937 | 1051
  Urological complications | 32 | 61
  Ocular involvement | 11 | 7
  Central nervous system involvement | 0 | 0
  Pneumonia/pulmonary abscess or necrotising involvement | 0 | 0
  Myocarditis | 0 | 0
  Diarrhoea: number analyzed (Participants) | 937 | 1051
  Diarrhoea | 12 | 15
  Any of the specified clinical complication | 321 | 424
Statistical Analysis 1: Comparison: PLWHIV and Mpox Coinfection vs HIV Negative PrEP Users With Mpox Infection; Statistical analysis of "Any of the specified clinical complications" measure; Test type: Superiority; p = 0.005, Chi-squared

3. Primary Outcome: Number of Hospitalisation Events
Description: Number of hospitalisations for clinical reasons only (i.e. not for precautionary measures or quarantine).
Time Frame: as for outcome 2
Measure: Number; unit: Events
Arm/Group | PLWHIV and Mpox Coinfection | HIV Negative PrEP Users With Mpox Infection
Number analyzed (Participants) | 946 | 1054
Events | 57 | 38
Statistical Analysis 1: Comparison: PLWHIV and Mpox Coinfection vs HIV Negative PrEP Users With Mpox Infection; Test type: Superiority; p = 0.011, Chi-squared

4. Primary Outcome: Death
Description: Number of any Mpox related mortality observed during the 3 month observation period
Time Frame: From date of disease onset (first symptom) until date of death related to Mpox (up to 3 months)
Measure: Count of Participants; unit: Participants
Arm/Group | PLWHIV and Mpox Coinfection | HIV Negative PrEP Users With Mpox Infection
Number analyzed (Participants) | 946 | 1054
Participants | 0 | 0

5. Primary Outcome: Differences in Mpox Lesion Severity (the Clinical Manifestation) in PLWHIV and PrEP Users
Description: The severity of lesions will be determined based on the peak/maximum severity score over the observation period. Lesion severity will be classified ordinally as follows:
  * Not presenting with skin lesions (0 skin lesions)
  * Mild (1-24 lesions)
  * Moderate (25-99 skin lesions)
  * Severe (100-250 skin lesions)
  * Very severe (>250 skin lesions) Individuals with severe or very severe lesions (ie, ≥100 skin lesions) will be classified as having "severe lesions".
Time Frame: as for outcome 2
Measure: Number; unit: participants
Arm/Group | PLWHIV and Mpox Coinfection | HIV Negative PrEP Users With Mpox Infection
Number analyzed (Participants) | 946 | 1054
participants
  Not presenting with skin lesions | 36 | 61
  Mild | 676 | 805
  Moderate | 48 | 38
  Severe | 5 | 2
  Very severe | 1 | 0
  Unknown number of lesions | 180 | 148
Statistical Analysis 1: Comparison: PLWHIV and Mpox Coinfection vs HIV Negative PrEP Users With Mpox Infection; Statistical analysis relates to "not presenting with skin lesions" measure; Test type: Superiority; p = 0.002, Chi-squared

6. Primary Outcome: Differences in the Clinical Manifestation of Mpox in PLWHIV and PrEP Users by Site of Lesions
Description: Differences in the clinical manifestation of Mpox in PLWHIV and PrEP users by site of lesions. Site of lesions include genital (vulva/vaginal mucosa/penis/pubic area), ano-rectal/perianal, oral mucosa (lips/gums/oral/pharynx), face, trunk (chest/torso/abdomen/back) and limbs (arms/forearms/legs/hands/feet).
Time Frame: as for outcome 2
Population: Site of lesion data was not available for all participants due to the retrospective data collection in this study.
Measure: Number; unit: participants
Arm/Group | PLWHIV and Mpox Coinfection | HIV Negative PrEP Users With Mpox Infection
Number analyzed (Participants) | 896 | 976
participants
  Genital (vulva/vaginal mucosa/penis/pubic area) | 425 | 565
  Ano-rectal/perianal: number analyzed (Participants) | 894 | 973
  Ano-rectal/perianal | 454 | 409
  Oral mucosa (lips/gums/oral/pharynx): number analyzed (Participants) | 889 | 972
  Oral mucosa (lips/gums/oral/pharynx) | 149 | 133
  Face: number analyzed (Participants) | 890 | 971
  Face | 267 | 284
  Trunk (chest/torso/abdomen/back): number analyzed (Participants) | 889 | 970
  Trunk (chest/torso/abdomen/back) | 353 | 293
  Limbs (arms/forearms/legs/hands/feet): number analyzed (Participants) | 893 | 970
  Limbs (arms/forearms/legs/hands/feet) | 416 | 444

7. Primary Outcome: Differences in the Clinical Manifestation of Mpox in PLWHIV and PrEP Users by Severity Indicators
Description: Presence of severity indicators, below, was assessed in PLWHIV and PrEP Users with Mpox
  * Significant lower respiratory symptoms
  * Confusion/encephalitis,
  * Other complications (e.g. secondary bacterial infection, sepsis)
  * Widely disseminated lesions and very many in number (≥100)
  * Suspected infection of the cornea
  * Severe, refractory pain from lesions requiring hospitalisation
  * Lesions associated with complications due to pain or swelling
Time Frame: as for outcome 2
Population: Severity indicators were not available for all participants due to the retrospective nature of this data collection study.
Measure: Number; unit: participants
Arm/Group | PLWHIV and Mpox Coinfection | HIV Negative PrEP Users With Mpox Infection
Number analyzed (Participants) | 938 | 1052
participants
  Significant lower respiratory symptoms: number analyzed (Participants) | 938 | 1051
  Significant lower respiratory symptoms | 1 | 1
  Confusion/Encephalitis: number analyzed (Participants) | 938 | 1051
  Confusion/Encephalitis | 0 | 0
  Other complications (eg, secondary bacterial infection): number analyzed (Participants) | 937 | 1049
  Other complications (eg, secondary bacterial infection) | 98 | 122
  Widely disseminated lesions and very many in number: number analyzed (Participants) | 933 | 1045
  Widely disseminated lesions and very many in number | 5 | 2
  Suspected infection of the cornea: number analyzed (Participants) | 938 | 1051
  Suspected infection of the cornea | 8 | 5
  Severe, refractory pain from lesions requiring hospitalisation | 19 | 3
  Lesions associated with complications due to pain: number analyzed (Participants) | 937 | 1051
  Lesions associated with complications due to pain | 27 | 34

8. Primary Outcome: Differences in the NEWS2 Score ≥5 (Severity Indicator) in PLWHIV and PrEP Users With Mpox
Description: National Early Warning Score [NEWS] 2 score of ≥5 was reported for PLWHIV and PrEP Users with Mpox.
  NEWS2 is a summary score of six physiological parameters (respiratory rate, oxygen saturation, systolic blood pressure, heart rate, level of consciousness, temperature, and supplemental oxygen dependency) routinely recorded for inpatients. Each parameter is assigned a score between 0-3 based on how far it deviates from the normal range. These parameters are used to generate an aggregate severity score classified as low: aggregate score 0-4, low -medium/medium: score of 3 in any individual parameter/aggregate score 5-6,high: aggregate score 7 or more. Minimum scale score is 0, Maximum scale score is 20.
  A higher score indicates a greater clinical risk and worse outcome. A score ≥5 is a key threshold for urgent clinical review and signifies severe disease.
Time Frame: as for outcome 2
Population: NEWS2 score was not available for all participants due to the retrospective nature of this data collection study.
Measure: Number; unit: participants
Arm/Group | PLWHIV and Mpox Coinfection | HIV Negative PrEP Users With Mpox Infection
Number analyzed (Participants) | 630 | 440
participants | 1 | 0

9. Primary Outcome: Differences in the Drug Treatments of Mpox in PLWHIV and PrEP Users
Description: Differences in the drug treatments (clinical manifestation) of Mpox in PLWHIV and PrEP users
Time Frame: as for outcome 2
Population: Drug treatment for mpox data was not available for all participants. Due to the retrospective nature of this data collection study, only available data was collected for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | PLWHIV and Mpox Coinfection | HIV Negative PrEP Users With Mpox Infection
Number analyzed (Participants) | 942 | 1044
Participants
  Tecovirimat | 10 | 4
  Other antimicrobials or antivirals | 3 | 3
  Any drug treatment for mpox | 13 | 7
Statistical Analysis 1: Comparison: PLWHIV and Mpox Coinfection vs HIV Negative PrEP Users With Mpox Infection; Statistical analysis relates to "any drug treatment for mpox" measure; Test type: Superiority; p = 0.114, Chi-squared

10. Primary Outcome: Differences in the Drug Treatments for Complications of Mpox in PLWHIV and PrEP Users
Description: Differences in the drug treatments for complications of Mpox (secondary infections, bronchopneumonia, sepsis, encephalitis, and infection of the cornea with ensuing loss of vision) in PLWHIV and PrEP users
Time Frame: as for outcome 2
Population: Drug treatment for Mpox complications data was not available for all participants. Due to the retrospective nature of this data collection study, only available data was collected for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | PLWHIV and Mpox Coinfection | HIV Negative PrEP Users With Mpox Infection
Number analyzed (Participants) | 942 | 1043
Participants
  Any drug for complications | 292 | 409
  Antibiotics | 170 | 209
  Analgesia | 246 | 333
  Laxatives | 32 | 56
Statistical Analysis 1: Comparison: PLWHIV and Mpox Coinfection vs HIV Negative PrEP Users With Mpox Infection; Statistical analysis relates to "any drug for complications" measure; Test type: Superiority; p < 0.001, Chi-squared

11. Primary Outcome: Differences in the First Symptom at Onset of Mpox in PLWHIV and PrEP Users
Description: First symptom at Mpox onset including lesion onset, prodromal symptoms (e.g., fever, myalgia, etc), rectal pain or other symptoms.
Time Frame: Mpox onset
Population: First symptom at Mpox onset was not available/unknown for all participants due to the retrospective data collection in this study.
Measure: Number; unit: participants
Arm/Group | PLWHIV and Mpox Coinfection | HIV Negative PrEP Users With Mpox Infection
Number analyzed (Participants) | 946 | 1054
participants
  Lesion onset | 322 | 500
  Prodromal symptoms (eg, fever, myalgia, etc) | 425 | 327
  Rectal pain | 66 | 47
  Other | 76 | 72
  Unknown | 57 | 108
Statistical Analysis 1: Comparison: PLWHIV and Mpox Coinfection; Test type: Superiority — Statistical analysis relates to "lesion onset" measure; p < 0.001, Chi-squared

12. Primary Outcome: Mpox Transmission
Description: Differences between Mpox transmission characteristics in PLWHIV and PrEP users
Time Frame: Mpox onset
Measure: Number; unit: participants
Arm/Group | PLWHIV and Mpox Coinfection | HIV Negative PrEP Users With Mpox Infection
Number analyzed (Participants) | 946 | 1054
participants
  Recent travel to/living in endemic country or country with outbreak | 95 | 262
  No recent travel to/living in endemic country or country with outbreak | 777 | 701
  Unknown recent travel to/living in endemic country or country with outbreak | 74 | 91
  Contact with suspected, probable, or confirmed case | 173 | 126
  No contact with suspected, probable, or confirmed case | 211 | 153
  Unknown contact with suspected, probable, or confirmed case | 562 | 775
  Contact with infected animal | 0 | 0
  No contact with infected animal | 580 | 402
  Unknown contact with infected animal | 366 | 652

13. Primary Outcome: Mpox Transmission Characteristics
Description: Differences in days between symptom onset and positive PCR test between PLWHIV with mpox and PrEP Users with mpox
Time Frame: Mpox onset
Population: Days between symptom onset and positive PCR test data was not available for all participants due to the retrospective nature of this data collection study.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | PLWHIV and Mpox Coinfection | HIV Negative PrEP Users With Mpox Infection
Number analyzed (Participants) | 850 | 940
days | 6 [4 to 9] | 7 [5 to 10]

14. Primary Outcome: Risk Factors for Mpox Outcomes
Description: Predicted risk factors (chronic kidney or liver disease, diabetes, lymphoma, AIDS defining condition, mental health condition, other comorbidities, and immunosuppression) will be analysed for presence or absence of severe mpox lesions (≥100 skin lesions)
Time Frame: as for outcome 2
Population: Severe lesion endpoint data was not available for all participants due to the retrospective nature of this data collection study. No events occurred in some groups and were therefore not included in this analysis.
Measure: Number; unit: participants
Groups:
- All Participants in Risk Predictor Category With Severe Mpox Lesions Present; All Participants in Risk Predictor Category With Severe Mpox Lesions Absent: PLWHIV and PrEP (Pre-exposure prophylaxis) users who are at least 18 years of age, with confirmed MPX infection by documented, positive result on PCR testing of lesions from 1st May 2022 to 1st December 2023
Arm/Group | All Participants in Risk Predictor Category With Severe Mpox Lesions Present | All Participants in Risk Predictor Category With Severe Mpox Lesions Absent
Number analyzed (Participants) | 1672 | 1672
participants
  Patient group -PLWHIV: number analyzed (Participants) | 766 | 766
  Patient group -PLWHIV | 6 | 760
  Patient group -PrEP users: number analyzed (Participants) | 906 | 906
  Patient group -PrEP users | 2 | 904
  Age <30: number analyzed (Participants) | 269 | 269
  Age <30 | 0 | 269
  Age 30-40: number analyzed (Participants) | 796 | 796
  Age 30-40 | 6 | 790
  Age > 40: number analyzed (Participants) | 607 | 607
  Age > 40 | 2 | 605
  Chronic kidney or liver disease: number analyzed (Participants) | 37 | 37
  Chronic kidney or liver disease | 2 | 35
  AIDS defining condition: number analyzed (Participants) | 308 | 308
  AIDS defining condition | 1 | 307
  Mental health condition: number analyzed (Participants) | 86 | 86
  Mental health condition | 1 | 85
  Immunosuppression: number analyzed (Participants) | 73 | 73
  Immunosuppression | 1 | 72
  Multiple sexual partners: number analyzed (Participants) | 1090 | 1090
  Multiple sexual partners | 2 | 1088
  Orthopoxvirus vaccination: number analyzed (Participants) | 92 | 92
  Orthopoxvirus vaccination | 1 | 91

15. Primary Outcome: Risk Factors for Mpox Outcomes for PLWHIV
Description: Risk factors (CD4 count) for severe mpox lesions (≥100 skin lesions) for PLWHIV
Time Frame: From date of disease onset (first symptom) until date of clinical resolution e.g. lesion resolution, hospital discharge or death(up to 3 months)
Population: CD4 data was not available for all participants due to the retrospective nature of this data collection study.
Measure: Mean (Standard Deviation); unit: cells/mm^3
Groups:
- PLWHIV With CD4 Count and Severe Mpox Lesions Present; PLWHIV With CD4 Count and Severe Mpox Lesions Absent: PLWHIV who are at least 18 years of age, with confirmed MPX infection by documented, positive result on PCR testing of lesions from 1st May 2022 to 1st December 2023
Arm/Group | PLWHIV With CD4 Count and Severe Mpox Lesions Present | PLWHIV With CD4 Count and Severe Mpox Lesions Absent
Number analyzed (Participants) | 5 | 649
cells/mm^3 | 680 (513) | 683 (338)

16. Secondary Outcome: Prevalence of Mpox During the Study Period
Description: The number of mpox patients attending sites as a percentage of total number of patients the sites have seen over a set period of time (from first Mpox patient to last Mpox patient)
Time Frame: 1st May 2022 to 1st December 2023
Population: All patient data was not available at 2 sites, Hospital Clinic Barcelona and EECE Warsaw, and are excluded from this analysis.
Measure: Number (95% Confidence Interval); unit: percentage of mpox cases
Groups:
- All Patients: Total number of patients evaluated at clinical sites 1st May 2022 to 1st December 2023.
Arm/Group | All Patients
Number analyzed (Participants) | 468845
percentage of mpox cases
  Chelsea and Westminster | 0.34 [0.32 to 0.36]
  Hospital Germans Trias i Pujol | 0.85 [0.76 to 0.94]
  Hospital San Carlos | 0.99 [0.92 to 1.07]
  Hospital Vall d'Hebron | 2.90 [2.63 to 3.19]
  Hospital La Paz | 1.54 [1.37 to 1.73]
  Hospital Bichat Claude-Bernard | 3.07 [2.90 to 3.26]
  Hospital Pitié Salpêtrière | 1.48 [1.33 to 1.64]

17. Secondary Outcome: Length of Stay in Hospital
Description: The length of stay in hospital for inpatients treated for Mpox. In the case of multiple hospitalisations, the sum of the length of all stays will be analysed.
Time Frame: From date of hospital admission for Mpox until date of hospital discharge (up to 3 months)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | PLWHIV and Mpox Coinfection | HIV Negative PrEP Users With Mpox Infection
Number analyzed (Participants) | 57 | 38
days | 6 [3 to 10] | 6 [2 to 9]

18. Secondary Outcome: Time to Lesion Resolution (if Known)
Description: The estimate the time to lesion resolution for participants with at least one lesion during the observation period and with a known date of lesion resolution will be included.
Time Frame: From date of disease onset (first symptom) until date of lesion resolution (up to 3 months)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | PLWHIV and Mpox Coinfection | HIV Negative PrEP Users With Mpox Infection
Number analyzed (Participants) | 241 | 162
days | 18 [13 to 24] | 17 [14 to 23]

ADVERSE EVENTS:
Time Frame: From date of disease onset/first symptom, D0, until date of clinical resolution e.g. lesion resolution, hospital discharge or death (up to 3 months) D90
Description: Adverse events were not assessed for this study, only deaths and hospitalisations were collected.
Arm/Group | PLWHIV and Mpox Coinfection | HIV Negative PrEP Users With Mpox Infection
All-Cause Mortality (participants affected / at risk) | 0/946 | 0/1054
Serious Adverse Events (participants affected / at risk) | 57/946 | 38/1054
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PLWHIV and Mpox Coinfection (N=946) | HIV Negative PrEP Users With Mpox Infection (N=1054)
Hospitalisation (General disorders) | 57 | 38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-01): https://cdn.clinicaltrials.gov/large-docs/27/NCT05965427/Prot_SAP_000.pdf